CLINICAL TRIAL: NCT03483194
Title: Therapeutic Virtual Reality : Impact on the Management of Pain and Anxiety Related to Hematology Care
Brief Title: Therapeutic Virtual Reality : Impact on the Management of Pain and Anxiety Related to Hematology Care (REVEH)
Acronym: REVEH
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Weprom (Other)
Collaborators: L'effet Papillon (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: WP-2017-01; 2017-A02701-52 (Other: French Health Products Safety Agency)
Record Dates: First submitted 2018-03-15; First posted 2018-03-30 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2019-07

CONDITIONS: Hematologic Neoplasms
Keywords: Therapeutic Virtual Reality; Pain related medical procedure management; Anxiety management; Osteo-medullary biopsy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — kalinox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kalinox® (Active Comparator): The included patients in this group will have, during the intervention, a local anesthesia by xylocaine® 10 mg / mL (1 bottle of 20 mL) in complement of a gas mixture composed of 50% Nitrous Oxide, 50% Oxygen (Kalinox®)
  Interventions: Drug: Kalinox
- Virtual Reality (Experimental): The included patients in this group will have, during the intervention, a local anesthesia by xylocaine® 10 mg / mL (1 bottle of 20 mL) in complement of a virtual reality (VR) session.
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — Bliss is a 3D Interactive application designed to meet the needs of escape and relaxation of people in isolation and / or stress and / or during painful care here osteo-medullary biopsy
  Other Names: Bliss
  Arms: Virtual Reality
Drug: Kalinox — Usually take care of by a gas mixture composed of 50% Nitrous Oxide, 50% Oxygen for the medical procedure (osteo-medullary biopsy)
  Other Names: Control
  Arms: Kalinox®

SUMMARY:
The management of hematological malignancies justifies the completion of a complete assessment before the start of treatment. This assessment includes imaging tests (computed tomography, position emission tomography, cavitary scintigraphy), biology and very often an exploration of the bone marrow by anterior or posterior iliac biopsy. Pains related to the disease (node compression, invasion of solid organs) are taken care of at the diagnosis and often relieved by the start of the specific treatment.

However, pain related to medical procedure is often overlooked and can lead to psychological trauma in some patients who may refuse to repeat these essential actions to assess the response to treatment.

Anxiety contributes to pain and various relaxation techniques have already proven their effectiveness. The goal of the protocol is to reduce the pain and anxiety associated with medical procedure by using virtual reality with a helmet proposed at the time of the gesture.

DETAILED DESCRIPTION:
Today, one third of the population suffers from anxiety and 20% of French people suffer from chronic pain. Many health situations or pathologies lead to difficult or painful care. The impact of drug solutions to relieve patients is often limited and more and more scientific studies are demonstrating the benefits of virtual reality to reduce pain, anxiety and addictions.

In 2011, following an experience of close to patient, a person created "l'Effet Papillon", a social enterprise that aims to create a concrete social impact in the lives of people with cancer, in situations of fragility or isolation and those who accompany them. Since 2011 the social enterprise has supported nearly 3,000 patients and today, the Butterfly Effect is a real partner of health actors by adopting a holistic approach to wellness in the face of disease and fragility.

Taking full advantage of the benefits of virtual reality that, used in medical settings, can reduce pain and anxiety, Bliss is a 3D Interactive application designed to meet the needs of escape and relaxation of people in isolation and / or or stress.

Bliss has been developed for and with patients in partnership with physicians, researchers and experts in virtual reality for therapeutic purposes.

Bliss offer a new tool for relaxation and well-being that relaxes and distracts users from moments of stress or anxiety.

The management of hematological malignancies justifies the completion of a complete assessment before the start of treatment. This assessment includes imaging tests (computed tomography, position emission tomography, cavitary scintigraphy), biology and very often an exploration of the bone marrow by anterior or posterior iliac biopsy. Pains related to the disease (node compression, invasion of solid organs) are taken care of at the diagnosis and often relieved by the start of the specific treatment.

However, pain related to medical procedure is often overlooked and can lead to psychological trauma in some patients who may refuse to repeat these essential actions to assess the response to treatment. Anxiety contributes to pain and various relaxation techniques have already proven their effectiveness.

During the osteo-medullary biopsy the patient will lie on his stomach with his hands positioned under the head. This position is the one recommended by the French Society of Hematology for an osteo-medullary biopsy.

The osteo-medullary biopsy remains independent of the object of the study and will be carried out according to the national recommendations.

For patients randomized to the "Standard" arm, the treatment will be the same as that proposed outside the study (a gas mixture composed of 50% Nitrous Oxide, 50% Oxygen + 1 bottle of xylocaine® 20 mL at the concentration of 10 mg / mL).

For randomized patients in the "Virtual Reality" arm, the VR session should begin 5 minutes before the start of the procedure (+ 1 bottle of Xylocaine® 20 mL at a concentration of 10 mg / mL). The VR session will last between 15 and 30 minutes depending on the speed programmed. The patient can continue the session if the gesture ends before the end of the virtual reality program.

The goal of the protocol is to reduce the pain and anxiety associated with medical procedure by using virtual reality with a helmet proposed at the time of the gesture.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with malignant haematological pathology
2. Patient who must have an osteo-medullary biopsy for diagnostic purposes
3. Age ≥ 18 years
4. Performance Status < 3
5. Patient with no pelvic bone pain before inclusion
6. Patient with normal coagulation balance (TP, Activated Partial Thromboplastin Time, fibrin) and platelet count> 50 G / L
7. Patient affiliated to the social security scheme
8. Patient giving written consent before any specific procedure related to the study

Exclusion Criteria:

1. Patient regularly taking antalgic treatments from stage 2 or 3
2. Patient with congenital coagulation disorder or acquired or taking anticoagulant therapy such as: fluindione, acenocoumarol, warfarin, dabigatran, apixaban or rivaroxaban
3. Contraindication to a gas mixture composed of 50% Nitrous Oxide, 50% Oxygen administration: true allergy, severe respiratory failure requiring continuous oxygen therapy, emphysema, pneumothorax, history of air embolism or diving accident, epilepsy or uncontrolled neurological disorder, unsubstituted vitamin deficiency B12 and folic acid, abdominal gas distension
4. Any contraindication to the use of the headset: pacemaker or other implanted medical device
5. Pregnancy or breastfeeding
6. Persons deprived of liberty, under guardianship or under guardianship
7. Dementia, mental impairment or psychiatric condition that may compromise patient informed consent and / or protocol compliance and follow-up of the trial
8. Patient unable to undergo protocol monitoring for psychological, social, family or geographical reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-06-19 (Actual)

PRIMARY OUTCOMES:
Assessment of pain | Fifteen minutes after the osteo-medullary biopsy
  Pain will be evaluated by Visual Analog Scale (0 = no pain at 10 = worst possible pain).

SECONDARY OUTCOMES:
Assessment of tolerance | During or within fifteen minutes after the osteo-medullary biopsy
  Quotation of nausea, dizziness or headache according to CTCAE
Assessment of the anxiety by specific questionnaire | Fifteen minutes after the osteo-medullary biopsy
  Anxiety will be evaluated by Inventory of situational anxiety and anxiety trait (IASTA scale)
Assessment of the anxiety by blood pressure measurement | Fifteen minutes after the osteo-medullary biopsy
  Anxiety will be evaluated by bood pressure measurement
Assessment of the fear of pain by questionnaire | Assessment at Baseline
  Fear of pain will be evaluated by a specific questionnaire
Assessment of the fear of pain by Visual Analog Scale | Assessment at Baseline
  Fear of pain will be evaluated by a Visual Analog Scale (0 = no pain at 10 = worst possible pain).
Assessment of residual pain | One month after the osteo-medullary biopsy
  Pain will be evaluated by Visual Analog Scale (0 = no pain at 10 = worst possible pain).
Assessment of investigator's satisfaction | Fifteen minutes after the osteo-medullary biopsy
  Satisfaction will be evaluated by a questionnaire for investigators
Assessment of patient's satisfaction | Fifteen minutes after the osteo-medullary biopsy
  Satisfaction will be evaluated by a questionnaire for patients
Assessment of nurse's satisfaction | Fifteen minutes after the osteo-medullary biopsy
  Satisfaction will be evaluated by a questionnaire for nurses
Assessment of drug consumption related to the osteo-medullary biopsy (Xylocaine) | During the osteo-medullary biopsy
  Drug consumption related to medical procedure will be evaluated by the number of bottle of xylocaine® (bottle of 20 mL, concentration of 10mg/mL) used
Assessment of drug consumption related to the osteo-medullary biopsy (Kalinox) | During the osteo-medullary biopsy
  Drug consumption related to medical procedure will be evaluated by the duration of exposure of a gas mixture composed of 50% Nitrous Oxide, 50% Oxygen (time in minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Katell LE DU, MD, Principal Investigator — Centre Jean Bernard - Le Mans
Locations (5):
- France (5):
  - SOL Clinique Sainte-Anne, Strasbourg, Alsace
  - Institut Bergonié, Bordeaux, Gironde
  - CHU Angers, Angers, Pays de Loire
  - Centre Jean Bernard - Clinique Victor Hugo, Le Mans
  - HIA Bégin, Saint-Mandé, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le Du K, Septans AL, Maloisel F, Vanquaethem H, Schmitt A, Le Goff M, Clavert A, Zinger M, Bourgeois H, Dupuis O, Denis F, Bouchard S. A New Option for Pain Prevention Using a Therapeutic Virtual Reality Solution for Bone Marrow Biopsy (REVEH Trial): Open-Label, Randomized, Multicenter, Phase 3 Study. J Med Internet Res. 2023 Feb 15;25:e38619. doi: 10.2196/38619. PMID 36790852